CLINICAL TRIAL: NCT02742129
Title: Inorganic Nitrite Delivery to Improve Exercise Capacity in HFpEF
Acronym: INDIE-HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adrian Hernandez (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Aires Pharmaceuticals, Inc. (Industry); University of Vermont (Other); Université de Montréal (Other); Mayo Clinic (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, Professor of Medicine, DUMC; Director, Health Services and Outcomes Research, DCRI, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00071526; 5U10HL084904 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-04-18 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AIR001 Crossover to Placebo (Experimental): Phase 1: Participants will wear an accelerometer device daily but take no study drug for 14 days (washout period). On day 15, participants begin phase I study drug Nebulized Sodium Nitrite (AIR001) at 46 mg, at minimum of 4 hours apart, for 3 doses per day during the active portion of the participant's day. On day 22 participants increase study drug dose to 80 mg at the same frequency. Regardless of participant's ability to tolerate study drug or if the participant requires down-titration, participants will begin Phase 2. Phase 2: Is identical to Phase 1 except subject will be taking Placebo instead of AIR001.
  Interventions: Drug: Nebulized Sodium Nitrite; Drug: Placebo
- Placebo crossover to AIR001 (Placebo Comparator): Phase 1: Participants will wear an accelerometer device daily but take no study drug for 14 days (washout period). On day 15, participants begin phase I study drug (Placebo) at 46 mg, at minimum of 4 hours apart, for 3 doses per day during the active portion of the participant's day. On day 22 participants increase study drug dose to 80 mg at the same frequency. Regardless of participant's ability to tolerate study drug or if the participant requires down-titration, participants will begin Phase 2. Phase 2: Is identical to Phase 1 except subject will be taking Nebulized Sodium Nitrite (AIR001) instead of Placebo.
  Interventions: Drug: Nebulized Sodium Nitrite; Drug: Placebo

INTERVENTIONS:
Drug: Nebulized Sodium Nitrite — Inhaled, nebulized inorganic sodium nitrite vs. inhaled, nebulized placebo at a dose of 80 mg (or maximally tolerated dose) administered at a minimum of 4 hours apart, three times per day, during the active part of the day.
  Other Names: AIR001
Drug: Placebo — Inhaled, nebulized placebo vs. inhaled, nebulized inorganic sodium nitrite at a dose of 80 mg (or maximally tolerated dose) administered at a minimum of 4 hours apart, three times per day, during the active part of the day.

SUMMARY:
A randomized, double-blind, placebo-controlled crossover study to assess the effect of inorganic nitrite (NO2) on aerobic capacity (peak VO2) after four weeks of dosing. Approximately 100 participants will be enrolled in this 2*2 crossover study.

DETAILED DESCRIPTION:
Screen potential HFpEF patients for eligibility criteria and interest

Study Visit 1

• Initiate consent process and obtain written informed consent.

* Confirm with the participant that HF symptoms are the primary limitation to activity. If so, they proceed to CPET screening. If not, they are considered a screen fail.
* Obtain baseline bloods *- CBC, complete chemistry panel, biomarkers, biorepository and genetics (if agreed to participate) .
* Obtain CPET to verify patient eligibility peak VO2 ≤ 75% predicted and RER ≥ 1.0 (within 3 days prior to randomization) and establish baseline value.
* Qualifying patients perform additional baseline studies: history, assess NYHA class, physical exam, ECG, and KCCQ.
* Open label, single-dose run-in where patient receives maximal dose (80 mg) inhaled inorganic nitrite. Patients who do not tolerate the run-in are considered screen failures.
* Randomize qualifying patients.
* Dispense phase-1 study drug, nebulizers and accelerometers
* Participants take no study drug for two weeks (baseline).
* Participants take 46 mg study drug at a minimum of 4 hours apart, 3 times a day, during active part of the day for 7 days.
* Participants take 80 mg study drug at a minimum of 4 hours apart, 3 times a day, during active part of the day until returning for study visit 2 (at least 42 days but up to 49 days post-baseline visit).
* If side effects develop, participants can down-titrate to the previous dose.
* Participants are called frequently to reinforce study procedures and assess compliance.

Study Visit 2 (42-49 Days Post Study Visit 1)

• Participant holds study drug on day of visit.

* Review history, assess NYHA class, perform physical exam and KCCQ.
* Obtain blood draws ** - CBC, complete chemistry panel, biomarkers, biorepository (if agreed to participate).
* Obtain limited echocardiogram **.
* Perform CPET with Study Drug administered immediately before starting the CPET (primary endpoint).
* Change out accelerometer and dispense phase-2 study drug.
* Participants take no study drug for two weeks (washout).
* Participants take 46 mg study drug at a minimum of 4 hours apart, 3 times a day, during active part of the day for 7 days.
* Participants take 80 mg study drug at a minimum of 4 hours apart, 3 times a day, during active part of the day until returning for study visit 3 (at least 42 but up to 49 days after study visit 2).
* If side effects develop Participants can down-titrate to the previously tolerated dose.
* Participants are called frequently to reinforce study procedures and assess compliance.

Study Visit 3 (42-49 Days Post Study Visit 2) • Participant holds study drug on day of visit.

• Review history, assess NYHA class, perform physical exam and KCCQ

* Obtain blood draws** - CBC, complete chemistry panel, biomarkers, biorepository (if agreed to participate).
* Obtain limited echocardiogram**.
* Perform CPET with Study Drug administered immediately before starting the CPET (primary endpoint).
* Return accelerometer and phase-2 study drug.
* End of study drug (phase out).

Phone Visit and End of Study (14 Days Post Study Visit 3)

• A final phone visit is conducted to assess for adverse events.

*Visit 1: baseline blood draw needs to be completed prior to the CPET (if this is not feasible, then they cannot be obtained for at least 3 hours post the CPET and prior to the run-in test dose).

**Visit 2 and Visit 3: blood draws and limited echo need to be obtained prior to study drug administration (if this is not feasible, then it cannot be obtained for at least 3 hours post study drug administration)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Symptoms of dyspnea (NYHA class II-IV) without evidence of a non-cardiac or ischemic explanation for dyspnea
3. EF ≥ 50% as determined on imaging study within 12 months of enrollment with no change in clinical status suggesting potential for deterioration in systolic function
4. One of the following :

   * Previous hospitalization for HF with radiographic evidence (pulmonary venous hypertension, vascular congestion, interstitial edema, pleural effusion) of pulmonary congestion or
   * Catheterization documented elevated filling pressures at rest (PCWP ≥15 or LVEDP ≥18) or with exercise (PCWP ≥25) or
   * Elevated NT-proBNP (>400 pg/ml) or BNP(>200 pg/ml) or
   * Echo evidence of diastolic dysfunction/elevated filling pressures manifest by medial E/e' ratio≥15 and/or left atrial enlargement and chronic treatment with a loop diuretic for signs or symptoms of heart failure
5. Heart failure is primary factor limiting activity as indicated by answering # 2 to the following question:

My ability to be active is most limited by:

1. Joint, foot, leg, hip or back pain
2. Shortness of breath and/or fatigue and/or chest pain
3. Unsteadiness or dizziness
4. Lifestyle, weather, or I just don't like to be active

6. Peak VO2 ≤75% predicted with peak respiratory exchange ratio≥1.0 CPET Normal Values for Peak VO2* Criteria (ml/kg/min) 7. No chronic nitrate therapy or not using intermittent sublingual nitroglycerin (requirement for >1 SL nitroglycerin per week) within last 7 days 8. No daily use of phosphodiesterase 5 inhibitors or soluble guanylyl cyclase activators and willing to withhold prn use of phosphodiesterase 5 inhibitors for duration of study 9. Ambulatory (not wheelchair / scooter dependent) 10. Body size allows wearing of the accelerometer belt as confirmed by ability to comfortably fasten the test belt provided for the screening process (belt designed to fit persons with BMI 20-40 kg/m2 but belt may fit some persons outside this range) 11. Willingness to wear the accelerometer belt for the duration of the trial 12. Willingness to provide informed consent

Exclusion Criteria:

1. Recent (< 1 month) hospitalization for heart failure
2. Ongoing requirement for PDE5 inhibitor, organic nitrate or soluble guanylyl cyclase activators
3. Hemoglobin (Hgb) < 8.0 g/dl within 90 days prior to randomization
4. GFR < 20 ml/min/1.73 m2 within 90 days prior to randomization
5. Systolic blood pressure < 115 mmHg seated or < 90 mmHg standing just prior to test dose
6. Resting HR > 110 just prior to test dose
7. Previous adverse reaction to the study drug which necessitated withdrawal of therapy
8. Significant chronic obstructive pulmonary disease thought to contribute to dyspnea
9. Ischemia thought to contribute to dyspnea
10. Documentation of previous EF < 45%
11. Acute coronary syndrome within 3 months defined by electrocardiographic (ECG) changes and biomarkers of myocardial necrosis (e.g., troponin) in an appropriate clinical setting (chest discomfort or anginal equivalent)
12. PCI, coronary artery bypass grafting, or new biventricular pacing within past 3 months
13. Primary hypertrophic cardiomyopathy
14. Infiltrative cardiomyopathy (amyloid)
15. Constrictive pericarditis or tamponade
16. Active myocarditis
17. Complex congenital heart disease
18. Active collagen vascular disease
19. More than mild aortic or mitral stenosis
20. Intrinsic (prolapse, rheumatic) valve disease with moderate to severe or severe mitral, tricuspid or aortic regurgitation
21. Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.7 in the absence of anticoagulation treatment
22. Terminal illness (other than HF) with expected survival of less than 1 year
23. Regularly (> 1x per week) swims or does water aerobics
24. Enrollment or planned enrollment in another therapeutic clinical trial in next 3 months.
25. Inability to comply with planned study procedures
26. Pregnancy or breastfeeding mothers

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hernandez, MD, Principal Investigator — Duke Clinical Research Institute; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (20):
- United States (20):
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston V.A. Healthcare System, West Roxbury, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri Health System, Columbia, Missouri
  - V.A St. Louis Health Care System, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - The University of Vermont - Fletcher Allen Health Care, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
After study completion, and upon site request, site specific participant data will be shared upon site requests. Sites may share this data with participants according to their individual institution's Institutional Review Board (IRB) policy.

REFERENCES:
- [Derived] Reddy YNV, Rikhi A, Obokata M, Shah SJ, Lewis GD, AbouEzzedine OF, Dunlay S, McNulty S, Chakraborty H, Stevenson LW, Redfield MM, Borlaug BA. Quality of life in heart failure with preserved ejection fraction: importance of obesity, functional capacity, and physical inactivity. Eur J Heart Fail. 2020 Jun;22(6):1009-1018. doi: 10.1002/ejhf.1788. Epub 2020 Mar 9. PMID 32150314
- [Derived] Borlaug BA, Anstrom KJ, Lewis GD, Shah SJ, Levine JA, Koepp GA, Givertz MM, Felker GM, LeWinter MM, Mann DL, Margulies KB, Smith AL, Tang WHW, Whellan DJ, Chen HH, Davila-Roman VG, McNulty S, Desvigne-Nickens P, Hernandez AF, Braunwald E, Redfield MM; National Heart, Lung, and Blood Institute Heart Failure Clinical Research Network. Effect of Inorganic Nitrite vs Placebo on Exercise Capacity Among Patients With Heart Failure With Preserved Ejection Fraction: The INDIE-HFpEF Randomized Clinical Trial. JAMA. 2018 Nov 6;320(17):1764-1773. doi: 10.1001/jama.2018.14852. PMID 30398602
- [Derived] Reddy YNV, Lewis GD, Shah SJ, LeWinter M, Semigran M, Davila-Roman VG, Anstrom K, Hernandez A, Braunwald E, Redfield MM, Borlaug BA. INDIE-HFpEF (Inorganic Nitrite Delivery to Improve Exercise Capacity in Heart Failure With Preserved Ejection Fraction): Rationale and Design. Circ Heart Fail. 2017 May;10(5):e003862. doi: 10.1161/CIRCHEARTFAILURE.117.003862. PMID 28476756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a diagnosis of HFpEF are screened for entry criteria. Willing participants meeting entry criteria will be consented and questioned to confirm that HF symptoms are the primary limitation to activity.
Pre-assignment Details: All consented participants continuing to meet the screening criteria will undergo a baseline HFN study-specific CPET to confirm Peak VO2 ≤75% with peak respiratory exchange ratio ≥ 1.0. All subjects that fulfill the CPET and other inclusion criteria and none of the exclusion criteria will be randomized.
Period: Phase 1
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Started | 53 | 52
Completed | 51 | 50
Not Completed | 2 | 2
Period: Phase 2
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Started | 51 | 50
Completed | 50 | 48
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- AIR001 Crossover to Placebo: Phase 1: Participants will wear an accelerometer device daily but take no study drug for 14 days (washout period). On day 15, participants begin phase I study drug Nebulized Sodium Nitrite (AIR001) at 46 mg, at minimum of 4 hours apart, for 3 doses per day during the active portion of the participant's day. On day 22 participants increase study drug dose to 80 mg at the same frequency. Regardless of participant's ability to tolerate study drug or if the participant requires down-titration, participants will begin Phase 2. Phase 2: Is identical to Phase 1 except subject will be taking Placebo instead of AIR001.
  Nebulized Sodium Nitrite: Inhaled, nebulized inorganic sodium nitrite vs. inhaled, nebulized placebo at a dose of 80 mg (or maximally tolerated dose) administered at a minimum of 4 hours apart, three times per day, during the active part of the day. Placebo: Inhaled, nebulized placebo vs. inhaled, nebulized inorganic sodium nitrite at a dose of 80 mg (or maximally to
- Placebo Crossover to AIR001: Phase 1: Participants will wear an accelerometer device daily but take no study drug for 14 days (washout period). On day 15, participants begin phase I study drug (Placebo) at 46 mg, at minimum of 4 hours apart, for 3 doses per day during the active portion of the participant's day. On day 22 participants increase study drug dose to 80 mg at the same frequency. Regardless of participant's ability to tolerate study drug or if the participant requires down-titration, participants will begin Phase 2. Phase 2: Is identical to Phase 1 except subject will be taking Nebulized Sodium Nitrite (AIR001) instead of Placebo.
  Nebulized Sodium Nitrite: Inhaled, nebulized inorganic sodium nitrite vs. inhaled, nebulized placebo at a dose of 80 mg (or maximally tolerated dose) administered at a minimum of 4 hours apart, three times per day, during the active part of the day. Placebo: Inhaled, nebulized placebo vs. inhaled, nebulized inorganic sodium nitrite at a dose of 80 mg (or maximally
- Total: Total of all reporting groups
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001 | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.5) | 67.5 (11.6) | 67.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 23 | 59
  Male | 17 | 29 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 53 | 51 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 47 | 45 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak VO2
Description: The primary endpoint will be the peak VO2 after 4 weeks treatment with inorganic nitrite as compared to the peak VO2 after 4 weeks treatment with placebo as assessed by cardiopulmonary exercise testing (CPET) performed at peak drug levels.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
ml/kg/min
  Phase 1: number analyzed (Participants) | 49 | 48
  Phase 1 | 13.4 (3.2) | 13.8 (3.8)
  Phase 2: number analyzed (Participants) | 49 | 45
  Phase 2 | 13.7 (3.0) | 13.6 (3.6)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — The statistical analysis compared the patient level data collected during the AIR001 period to the data collected during the placebo period. The Outcome Measure data is displaying the data as collected during each study phase and is combined together based upon expected treatment assignment for analysis; p = 0.2650, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.56 to 0.16]

2. Secondary Outcome: Average Arbitrary Accelerometer Units (AAU)
Description: Average arbitrary accelerometer units (AAU) during at least 14 days and up to 21 days of the maximally tolerated dose of study drug (from 28 days post Study Visit 1 until Study Visit 2 and from 28 days post Study Visit 2 until Study Visit 3). An arbitrary accelerometer unit is calculated within the accelerometer device that is worn by the patient and represents level of activity based upon patient movement. Higher values indicate more movement. Zero indicates no movement.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: accelerometry units
Groups:
- AIR001 Crossover to Placebo: Phase 1: Participants will wear an accelerometer device daily but take no study drug for 14 days (washout period). On day 15, participants begin phase I study drug (AIR001) at 46 mg, at minimum of 4 hours apart, for 3 doses per day during the active portion of the participant's day. On day 22 participants increase study drug dose to 80 mg at the same frequency. Regardless of participant's ability to tolerate study drug or if the participant requires down-titration, participants will begin Phase 2. Phase 2: Is identical to Phase 1 except subject will be taking Placebo instead of AIR001.
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
accelerometry units
  Phase 1: number analyzed (Participants) | 49 | 47
  Phase 1 | 5692 (2886) | 5341 (3115)
  Phase 2: number analyzed (Participants) | 41 | 46
  Phase 2 | 5688 (2950) | 5289 (2976)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9069, Mixed Models Analysis; Mean Difference (Final Values) = -14.68, 95% CI 2-sided [-263.65 to 234.29]

3. Secondary Outcome: Medial E/e' Ratio as Measured by Echocardiography Core Lab
Description: To evaluate whether AIR001 improves Medial E/e' ratio (the ratio between early mitral inflow velocity and mitral annular early diastolic velocity for diastolic evaluation) in comparison to placebo.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
ratio
  Phase 1: number analyzed (Participants) | 46 | 44
  Phase 1 | 15.4 (8.3) | 18.3 (11.8)
  Phase 2: number analyzed (Participants) | 47 | 46
  Phase 2 | 15.0 (7.3) | 17.4 (11.1)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9338, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.16 to 1.27]

4. Secondary Outcome: Left Atrial Volume Index as Measured by Echocardiography
Description: To evaluate whether AIR001 improves Left atrial volume index in comparison to placebo.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
ml/m^2
  Phase 1: number analyzed (Participants) | 44 | 37
  Phase 1 | 36.3 (16.5) | 40.1 (20.6)
  Phase 2: number analyzed (Participants) | 40 | 40
  Phase 2 | 37.2 (13.9) | 39.1 (20.4)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8151, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-2.79 to 2.20]

5. Secondary Outcome: Pulmonary Artery Systolic Pressure as Measured by Echocardiography
Description: To evaluate whether AIR001 improves pulmonary artery systolic pressure in comparison to placebo.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
mmHg
  Phase 1: number analyzed (Participants) | 38 | 36
  Phase 1 | 38.2 (9.7) | 39.6 (13.5)
  Phase 2: number analyzed (Participants) | 32 | 38
  Phase 2 | 35.0 (7.3) | 37.3 (9.2)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4658, Mixed Models Analysis; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-1.41 to 3.05]

6. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Score
Description: To evaluate whether AR001 improves quality of life in comparison to placebo. The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific patient-reported outcomes measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Symptom Burden, Symptom Stability, Physical Limitation, Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scale and summary scores range between 0 and 100, with higher scores indicating better health status (eg, better functioning, fewer symptoms, better quality of life). Higher values of the overall KCCQ score are considered to be better than lower values.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
units on a scale
  Phase 1: number analyzed (Participants) | 50 | 49
  Phase 1 | 65.6 (18.8) | 59.8 (18.4)
  Phase 2: number analyzed (Participants) | 49 | 48
  Phase 2 | 64.1 (18.4) | 59.4 (21.1)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3902, Mixed Models Analysis; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [-1.37 to 3.49]

7. Secondary Outcome: N-terminal Pro-B-type Natriuretic Peptide Level (NT-proBNP)
Description: Evaluate whether AIR001 improves natriuretic peptide levels in comparison to placebo
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
pg/mL
  Phase 1: number analyzed (Participants) | 48 | 49
  Phase 1 | 494.8 (542.3) | 550.4 (746.5)
  Phase 2: number analyzed (Participants) | 47 | 48
  Phase 2 | 513.9 (606.0) | 545.2 (784.5)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7404, Mixed Models Analysis; Mean Difference (Final Values) = 10.69, 95% CI 2-sided [-53.21 to 74.6]

8. Secondary Outcome: NYHA (New York Heart Association) Class
Description: To evaluate whether AR001 improves NYHA Class in comparison to placebo. NYHA class was measured at the end of each phase. The site physician evaluated the patient based upon the criteria for NYHA class I-IV used by the American Heart Association. NYHA functional classification provides a way of classifying the extent of heart failure. Class I (least severe): No limitation of physical activity; Class II: Slight limitation of physical activity; Class III: Marked limitation of physical activity; Class IV (most severe): Unable to carry on any physical activity without discomfort.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
Participants
  Phase 1: number analyzed (Participants) | 49 | 49
  Phase 1: I | 1 | 0
  Phase 1: II | 21 | 29
  Phase 1: III | 26 | 20
  Phase 1: IV | 1 | 0
  Phase 2: number analyzed (Participants) | 49 | 48
  Phase 2: I | 0 | 1
  Phase 2: II | 24 | 22
  Phase 2: III | 24 | 25
  Phase 2: IV | 1 | 0
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4282, Mixed Models Analysis; Median Difference (Final Values) = 0.05, 95% CI 2-sided [-0.08 to 0.18]

9. Secondary Outcome: Patient Preference for AIR001 Treatment at the End of Study
Description: Self-reported participant preference for study period 1 (Phase 1) vs. study period 2 (Phase 2)
Time Frame: End of Phase 2
Population: All randomized patients with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 48 | 47
Participants
  Phase 1 Patient Felt Better | 23 | 15
  Phase 2 Patient Felt Better | 17 | 20
  No Preference | 8 | 12

10. Secondary Outcome: VE/VCO2 Slope (Ventilatory Efficiency) as Provided by Cardiopulmonary Exercise Testing Core Lab
Description: To evaluate whether ARI001 in comparison to placebo improves ventilator efficiency as measured by Slope of Ve/VCO2 during study drug administration. The Ve/VCO2 slope is defined as the slope of the linear relationship between ventilation and carbon dioxide output and is a measure of the velocity.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
unitless
  Phase 1: number analyzed (Participants) | 49 | 49
  Phase 1 | 31.8 (5.7) | 33.9 (6.9)
  Phase 2: number analyzed (Participants) | 48 | 45
  Phase 2 | 32.1 (6.0) | 33.6 (7.3)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1067, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.08 to 0.11]

11. Secondary Outcome: VO2 at Ventilatory Threshold (Submaximal Exercise Capacity) as Provided by Cardiopulmonary Exercise Testing Core Lab
Description: To evaluate whether ARI001 in comparison to placebo improves submaximal exercise capacity as measured by VO2 (rate of oxygen consumption measured during incremental exercise) at ventilatory threshold during study drug administration.
Time Frame: End of Phase 1 & End of Phase 2
Population: All patients randomized.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | AIR001 Crossover to Placebo | Placebo Crossover to AIR001
Number analyzed (Participants) | 53 | 52
ml/min
  Phase 1: number analyzed (Participants) | 47 | 45
  Phase 1 | 7.8 (1.6) | 8.0 (1.9)
  Phase 2: number analyzed (Participants) | 47 | 43
  Phase 2 | 7.9 (1.6) | 7.8 (1.7)
Statistical Analysis 1: Comparison: AIR001 Crossover to Placebo vs Placebo Crossover to AIR001; The mixed models used to generate the p-values included all patients, including those with incomplete data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4411, Mixed Models Analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.37 to 0.16]

ADVERSE EVENTS:
Time Frame: Consent to 2 weeks post end of Phase 2
Description: Per protocol, all AEs/SAEs were collected except for anticipated, disease-related events in patients with HF with preserved EF. If a patient stopped participation in the study for any reason prior to the beginning of a study phase, that patient would not be included in the denominator for the treatment received in the period that was missed.
Groups:
- AIR001: Time period in which patient received AIR001 plus 2 weeks regardless of study phase.
- Placebo: Time period in which patient received placebo plus 2 weeks regardless of study phase.
Arm/Group | AIR001 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/103 | 0/102
Serious Adverse Events (participants affected / at risk) | 5/103 | 4/102
Other Adverse Events (participants affected / at risk) | 79/103 | 51/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIR001 (N=103) | Placebo (N=102)
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIR001 (N=103) | Placebo (N=102)
Nausea (Gastrointestinal disorders) | 6 | 1
Fatigue (General disorders) | 6 | 3
Dizziness (Nervous system disorders) | 17 | 19
Headache (Nervous system disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 10
dsypnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Chest discomfort (General disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT02742129/SAP_000.pdf
  • Study Protocol (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT02742129/Prot_001.pdf